CLINICAL TRIAL: NCT03865095
Title: Muscle Mass Loss in Critically Ill and Its Risk Factors. A Prospective Observational Study.
Brief Title: Muscle Mass Loss in Critically Ill Patients.
Acronym: MUSIC
Status: Completed | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT0012019
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Muscle Loss
Keywords: Critical Care; Muscle loss; Rectus femoris cross sectional area; Muscle ultrasound
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to describe the change in muscle mass in critically ill patients. The study will examine rectus femoris cross sectional area with ultrasound and identify risk factors of this changes.

DETAILED DESCRIPTION:
The study will commence following the Approval by The Ethics Research Committee. All patients admitted to our ICU from the 1st of March 2019 to the 31st of August 2019 will be enrolled after fulfilling the inclusion criteria and in the absence of any exclusion criteria. Informed consent will be requested. Ultrasound measurement of rectus femoris cross sectional area will be performed in first 24 hours after admission to ICU.

Study data will be entered in study form. The ultrasound measurement will be repeated on day 7 of hospitalisation.

Changes in rectus femoris cross sectional area and potential risk factors will be analysed. The length of ICU length of stay and 28-day mortality will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* mechanical ventilation expected for at least 48 hours

Exclusion Criteria:

* Clinical Frailty Score above 7 prior admission
* neuromuscular disease in previous medical history
* amputated lower extremities
* trauma of lower extremities involving tights
* age under 18 years
* inability to perform ultrasound examination
* death or discharge prior completion of protocol
* full verticalization prior completion of protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients admitted to intensive care unit with suspect length of artificial ventilation more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Muscle mass loss | 7 days
  Change in cross sectional area of rectus femoris muscle estimated by ultrasound

SECONDARY OUTCOMES:
28 day mortality | 28 days after enrolment
  mortality 28 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, M.D., PhD., Study Chair — University Hospital Brno and Masaryk University
Locations (1):
- University Hospital Brno and Masaryk University Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hrdy O, Vrbica K, Kovar M, Korbicka T, Stepanova R, Gal R. Incidence of muscle wasting in the critically ill: a prospective observational cohort study. Sci Rep. 2023 Jan 13;13(1):742. doi: 10.1038/s41598-023-28071-8. PMID 36639540